CLINICAL TRIAL: NCT05798611
Title: A Phase II, Open-label, Multi-center, Basket Study of the ATR Kinase Inhibitor ART0380 Administered Orally as Monotherapy to Patients With Biologically Selected Advanced or Metastatic Solid Tumors (ARTIST)
Brief Title: Study of ART0380 in Patients With Biologically Selected Solid Tumors
Acronym: ARTIST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision, not for reasons affecting the benefit-risk balance.
Sponsor: Artios Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART0380C004; 2023-504153-12 (EudraCT Number)
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Recurrent Endometrial Cancer; Metastatic Cancer
Keywords: Solid Tumors; Monotherapy; Cancer cell; Oral anti-cancer
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 [ART0380 monotherapy (endometrial cancer patients)] (Experimental): Patients with persistent or recurrent endometrial cancer (EC) will receive ART0380 monotherapy in one of two dose regimens for a 21-day cycle.
  Interventions: Drug: ART0380
- Arm 2 [ART0380 monotherapy (solid tumors patients)] (Experimental): Patients with advanced or metastatic solid tumors will receive ART0380 monotherapy in one of two dose regimens for a 21-day cycle.
  Interventions: Drug: ART0380

INTERVENTIONS:
Drug: ART0380 — Randomized patients will orally receive ART0380.

SUMMARY:
This interventional study will evaluate the efficacy and safety of ART0380 as monotherapy in patients whose tumors have a biology to predict for sensitivity to inhibition of Ataxia-Telangiectasia Mutated and Rad3-related protein kinase (ATR).

DETAILED DESCRIPTION:
ART0380 is being developed as an oral anti-cancer agent for the treatment of patients with cancers that have defects in deoxyribonucleic acid (DNA) repair.

The study will recruit selected patients with advanced or metastatic solid tumors, specifically:

* Patients with persistent or recurrent endometrial cancer (EC)
* Patients with advanced or metastatic solid tumors of any histology

Above patients will be randomized in a 1:1 ratio to one of two dose regimens of ART0380.

Safety will be evaluated on a quarterly basis, at a minimum. Patients may continue to receive ART0380 as long as they are continuing to derive benefit from treatment or until disease progression, withdrawal of consent, or until they experience unacceptable drug-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have discontinued all previous treatments for cancer for at least 21 days or 5 half-lives (not including palliative radiotherapy at focal sites), whichever is shorter. Palliative radiotherapy must have completed 1 week prior to start of study treatment.
* Resolution of all toxicities of prior therapy or surgical procedures to baseline or Grade 1 (except for hypothyroidism requiring medication, neuropathy, and alopecia, which must have resolved to Grade ≤2).
* Have adequate organ function.
* Patients of childbearing potential and patients with partners of childbearing potential are required to use highly effective contraception.
* Have an estimated life expectancy of ≥12 weeks, in the judgment of the investigator.
* Performance status of 0-1 on the Eastern Cooperative Oncology Group scale.
* Have a non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available.

Inclusion Criteria specific to each Arm

Inclusion Criteria for Arm 1 [ART0380 monotherapy (endometrial cancer patients)]

* Persistent or recurrent EC with biological selection.
* Patients should have received taxane/platinum chemotherapy unless contraindicated.
* Measurable disease.

Inclusion Criteria for Arm 2 [ART0380 monotherapy (solid tumors patients)]

* Advanced or metastatic solid cancers of any histology with biological selection.
* If a Programmed cell death protein-1 /Programmed death-ligand-1 inhibitor (e.g., pembrolizumab) is approved and available for the patient's cancer, the patient should have received such treatment before participating in this study.
* Radiologically evaluable disease.

Exclusion Criteria:

* Patients who are pregnant.
* Prior treatment with an inhibitor of ATR, WEE1, checkpoint kinase 1 or PKMYT1.
* Have a serious concomitant systemic disorder that would compromise the patient's ability to adhere to the protocol.
* Have ongoing interstitial lung disease or pneumonitis (whether symptomatic or asymptomatic).
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS) directed therapy shows no evidence of progression.
* Have any major gastrointestinal issues that could impact absorption of ART0380.
* Have a history of allergy or hypersensitivity to study drug components.
* Have a significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 12 weeks prior to enrollment.
* Patients who plan to father a child while in the study or within 16 weeks (5 months in France) after the last administration of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Until disease progression (Every 6 weeks from randomization Upto 2 Years)
  Objective Response Rate (ORR) is defined as the proportion of patients with a complete response (CR) or partial response (PR) to treatment according to Response evaluation criteria in solid tumors (RECIST v1.1).

SECONDARY OUTCOMES:
Number of patients with adverse events | From Cycle 1 (each Cycle is 21-day) Day 1 until 30-day follow-up visit (Upto 2 Years)
  To assess the safety and tolerability of ART0380 in patients with solid tumors.
Progression free survival (PFS) | Screening (≤28 days) Until disease progression (Every 6 weeks from randomization Upto 2 Years)
  The PFS is defined as the time from randomization until the earliest objective disease progression defined by RECIST v1.1 or Prostate Cancer Working Group 3 (PCWG-3) (for patients with prostate cancer in Arm 2) or death by any cause in the absence of progression, regardless of whether the patient withdraws from study medication or receives another anti-cancer therapy prior to progression.
Best overall response (BOR) | Screening (≤28 days) Until disease progression (Every 6 weeks from randomization Upto 2 Years)
  The best overall response is the best response (complete response, and partial response) recorded from the date of randomization for each patient until the progression or censoring date in the absence of progression.
Disease control rate (DCR) | Screening (≤28 days) Until disease progression (Every 6 weeks from randomization Upto 2 Years)
  To further explore the efficacy of ART0380 in patients with solid tumors enrolled in each of the biologically defined arms.
Duration of response (DOR) | Screening (≤28 days) Until disease progression or death (Every 6 weeks from randomization Upto 2 Years)
  The DOR will be defined for patients with a BOR of CR/PR, as the time from the date of first documented response until date of documented progression (by RECIST v1.1) or death in the absence of disease progression.
Change in tumor size | Screening (≤28 days) Until disease progression (Every 6 weeks from randomization Upto 2 Years)
  The best percentage change in tumor size from baseline will be determined for each patient, ie, the maximum reduction from baseline or the minimum increase from baseline in the absence of a reduction.
Overall survival (OS) | Screening (≤28 days) Until overall survival follow-up (Every 12 weeks until data cut-off)
  The OS is defined as the time from the randomization until death due to any cause.
Maximum plasma concentration (Cmax) | Pre-dose Cycle 1 day 1, 2, 15, 16, 17, 18, Cycle 2 day 1, Cycle 3 day 1 Upto 2 Years (Each Cycle is 21-days)
  To determine the Cmax of ART0380 following single oral dosing of ART0380 in patients with solid tumors enrolled in each of the biologically defined arms.
Half life (t1/2) | Pre-dose Cycle 1 days 1, 2, 15, 16, 17, 18, Cycle 2 day 1, Cycle 3 day 1 Upto 2 Years (Each Cycle is 21-days)
  To determine the t1/2 of ART0380 following single oral dosing of ART0380 in patients with solid tumors enrolled in each of the biologically defined arms.
Area under the plasma concentration-time curve from zero to infinity (AUC0-inf) | Pre-dose Cycle 1 days 1, 2, 15, 16, 17, 18, Cycle 2 day 1, Cycle 3 day 1 Upto 2 Years (Each Cycle is 21-days)
  To determine the AUC0-inf of ART0380 following single oral dosing of ART0380 in patients with solid tumors enrolled in each of the biologically defined arms.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (8):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - The University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Northwell Health R.J. Zuckerberg Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center (MSKCC) - Memorial Hospital - Oncology, New York, New York
  - University of Oklahoma/Sarah Cannon Research Institute, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
- France (5):
  - Institut de Cancérologie de l'Ouest, Angers, NAP
  - Centre Francois Baclesse - Service d'Oncologie médicale, Caen, NAP
  - Hopital Cochin Saint Vincent De Paul, Paris, NAP
  - Hopital Lyon Sud, Pierre-Bénite, NAP
  - Centre Hospitalier Universitaire De Poitiers, Poitiers, NAP
- Spain (2):
  - Hospital Universitario De Jaén, Jaén, Andalusia
  - Fundación Instituto Valenciano De Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No